CLINICAL TRIAL: NCT04685759
Title: Assessing the Non-inferiority of Virtual vs. In-person Concurrent Exercise Regimens in Patients Receiving Neoadjuvant Therapy Prior to Surgical Resection of a Primary GI Tumor
Brief Title: Exercise Regimens and Neoadjuvant Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited candidate pool
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jay Lohrey, Assistant Professor, Internal Medicine / Harold S. Simmons Comprehensive Cancer Center, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2020-0948
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cancer of Gastrointestinal Tract
Keywords: Exercise Therapy; Cancer of Gastrointestinal Tract; Neoadjuvant Therapies
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Exercise Protocol (IPEP) (Active Comparator): This group will receive exercise instruction and monitoring in-person from the certified Cancer Exercise Trainer (CET) in the gym facility at Moncrief Cancer Institute (MCI). Study participants will be scheduled for exercise sessions twice a week with the oncology exercise trainer.
  Interventions: Other: In-Person Exercise Protocol
- Virtual Exercise Protocol (VEP) (Experimental): This group will receive exercise instruction and monitoring from the CET via telehealth sessions at home. Study participants will be scheduled for exercise sessions twice a week with the oncology exercise trainer.
  Interventions: Other: Virtual Exercise Protocol

INTERVENTIONS:
Other: In-Person Exercise Protocol — Supervised aerobic, resistance, flexibility, balance, and agility exercises, which could include yoga for a total of approximately 75 minutes per in-person session.
  Arms: In-Person Exercise Protocol (IPEP)
Other: Virtual Exercise Protocol — Supervised aerobic, resistance, flexibility, balance, and agility exercises, which could include yoga for a total of approximately 75 minutes each virtual session. A TheraBand (resistance band) will be provided to patients in this group to be used for resistance and flexibility training.
  Arms: Virtual Exercise Protocol (VEP)

SUMMARY:
The purpose of this study is to assess the effectiveness of exercise therapy for patients undergoing neoadjuvant chemotherapy for primary gastrointestinal (GI) tract cancer, providing a reproducible exercise regimen designed to improve or preserve aerobic fitness, strength, and quality of life. In addition, this study will address shifts in healthcare delivery needed as a result of the coronavirus disease 2019 (COVID-19) pandemic, evaluating the effectiveness of telehealth instruction as a method for exercise therapy.

The study hypotheses are:

1. To evaluate the effectiveness of exercise therapy for cancer patients undergoing neoadjuvant treatment when delivered via telehealth, as compared to an in-person setting.
2. To assess stair test instrumentation, previously validated in a healthy population, as a measure to gauge health status in cancer patients undergoing neoadjuvant treatment.
3. To assess patient satisfaction with exercise therapy when delivered via telehealth, as compared to an in-person setting.

DETAILED DESCRIPTION:
After being informed about the study and potential risks and benefits, all patients meeting inclusion criteria who provide written informed consent will be randomized at the time of enrollment to one of two cohorts engaged in a standardized exercise regimen based on delivery method, either in-person or via telehealth. Patient function will be assessed using the Timed Up and Go (TUG) test; Stairs Test; which evaluates aerobic ability, resistance, agility, balance, and posture; and given a score on the Karnofsky Performance Status Scale. Patient quality of life will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) survey. Outcomes for the cohorts will be compared over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Primary language is either English or Spanish
* Primary cancer diagnosis of GI cancer
* Undergoing neoadjuvant chemotherapy prior to surgical resection.
* Patients are being treated by medical oncologist at Simmons Cancer Center at Moncrief Cancer Institute in Fort Worth

Exclusion Criteria:

* Patient has had systemic cancer treatment in the past year
* Patient initiated neoadjuvant chemotherapy treatment prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a primary GI tumor who complete neoadjuvant treatment and are cleared for surgical resection | Up to Week 12
  The primary efficacy endpoint is the proportion of patients who complete neoadjuvant treatment and surgical resection for a primary GI tumor. All individuals failing to achieve the success definition described above will be considered treatment failures. All individuals who drop out of the study or discontinue in the exercise program prior to completion of neoadjuvant chemotherapy (NAC) and surgical resection will be considered treatment failures. Patients will be evaluated for surgical resection at completion of NAC (Week 8-12).

SECONDARY OUTCOMES:
Change from baseline in aerobic ability, resistance, agility, balance, and posture as measured by the Timed Up and Go Test | Baseline prior to initial exercise therapy session, midpoint (Week 4, Up to Week 6), neoadjuvant chemotherapy completion prior to surgery (Week 8, Up to Week 16), and 30 days post-operative surgery for tumor removal.
  Analyses of change from baseline will be measured by the Timed Up and Go Test (TUG). Change from baseline measurement at 30 days post-op will be fit with terms for treatment group and the measurement at baseline. Values for subjects who do not undergo the final assessment will be imputed using the last recorded value.
  The TUG test is a validated measurement of patient agility and balance, in addition to assessing if patient is a fall risk. Patients will be timed in seconds on standing up from a seated position, walking to a 3 meter line, and returning to the chair in a seated position at their regular pace without assistance from another person.
  Reference values for ages 60-99 years range from 7.1-12.7 seconds, with additional cut-off values predictive of falls. Results correlate with gait speed, balance, functional level, the ability to go out, and can follow change over time.
Change from baseline in aerobic ability, resistance, agility, balance, and posture as measured by the Stair Test | Baseline prior to initial exercise therapy session, midpoint (Week 4, Up to Week 6), neoadjuvant chemotherapy completion prior to surgery (Week 8, Up to Week 16), and 30 days post-operative surgery for tumor removal.
  Analyses of change from baseline will be measured by the Stair Test. Change from baseline measurement at 30 days post-op will be fit with terms for treatment group and the measurement at baseline. Values for subjects who do not undergo the final assessment will be imputed using the last recorded value.
  The Stair test is a validated measurement of aerobic ability, resistance, agility, balance, and posture. Patients will be timed in seconds to climb 2 flights of stairs in a constant rhythm, one step at a time. Patients will not be allowed to stop at any point during the climb or use side railings for support. The cancer exercise trainer will accompany each subject to ensure protocol compliance and safety. Maximal oxygen intake (VO2max) will be calculated for each patient and compared against predicted VO2 calculations based on gender, age, BMI, and heart rate at end of the stair climb.
Change in patient function as measured by Karnosfky Performance Status Scale | Baseline prior to initial exercise therapy session, midpoint (Week 4, Up to Week 6), neoadjuvant chemotherapy completion prior to surgery (Week 8, Up to Week 16), and 30 days post-operative surgery for tumor removal.
  The Karnosfky Performance Status Scale measures the ability of cancer patients to perform ordinary tasks. Possible scores range from 0 to 100 by increments of 10, with higher scores indicating that patients are better able to carry out daily activities.
  Patient function will be assessed using the Timed Up and Go (TUG) test, Stairs Test, which evaluate patient's aerobic ability, resistance, agility, balance, and posture, as well as the Karnosfky Performance Status Scale. Patient quality of life will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) survey. All assessments will be completed at baseline, prior to the initial exercise therapy session, at midpoint, and at the final session prior to surgery, as well as 30 days post-surgery. Exercise therapy will be deemed effective by preventing a reduction to patient function and quality of life over the course of enrollment in the study.
Change in quality of life assessment | Baseline prior to initial exercise therapy session (Week 1), midpoint (Week 4, Up to Week 6), neoadjuvant chemotherapy completion prior to surgery (Week 8, Up to Week 16), and 30 days post-operative surgery for tumor removal (Week 13, Up to Week 17).
  Analyses of change from baseline for quality of life will be measured by the Functional Assessment of Cancer Therapy - General (FACT-G) survey. Change from baseline measurement at 30 days post-op will be fit with terms for treatment group and the measurement at baseline. Values for subjects who do not undergo the final assessment will be imputed using the last recorded value.
  The FACT-G survey measures patient quality of life. This validated survey contains 27 items measured by a 5 point Likert-type scale in 4 domains relevant to cancer patients: Physical, Social, Emotional, and Functional well-being.
  Possible scores range from 0 to 108, with higher scores indicating a better quality of life.

OTHER OUTCOMES:
Mean total Patient Satisfaction score of Telehealth Exercise Therapy | Immediately after administration of each exercise session
  The Virtual Exercise Protocol Satisfaction Survey Scale (VEPSS1) measures patient satisfaction with the service delivery method of the exercise intervention. This is a researcher-designed survey for use in this study. Possible scores range from 0 to 20, with higher scores indicating a better outcome. The VEPSS1 will be used for telehealth cohort only.
  Satisfaction will be summarize as a continuous score for the participant populations. Median and interquartile ranges of the score will be recorded. Differences in comprehension will be measured between the In-Person Exercise Protocol Satisfaction Survey Scale and the VEPSS1.
Mean total Patient Satisfaction score of In-Person Exercise Therapy | Immediately after administration of each exercise session
  The In-Person Exercise Protocol Satisfaction Survey Scale (IPEPSS1) measures patient satisfaction with the in-person service delivery method of the exercise intervention. This is a researcher-designed survey for use in this study. Possible scores range from 0 to 20, with higher scores indicating a better outcome. The IPEPSS1 will be used for in-person exercise cohort only.
  Satisfaction will be summarize as a continuous score for the participant populations. Median and interquartile ranges of the score will be recorded. Differences in comprehension will be measured between the IPEPSS1 and the VEPSS1.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Lohrey, Principal Investigator — Jay.Lohrey@UTSouthwestern.edu
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Moncrief Cancer Institute, Fort Worth, Texas
  - UT Southwestern Simmons Comprehensive Cancer Center - Fort Worth, Fort Worth, Texas